CLINICAL TRIAL: NCT07245888
Title: Endotyping of Ventilator-associated Pneumonia With Proteomics on Bronchoalveolar Lavage for Improved Diagnosis, the ClusterVAP Study
Brief Title: ClusterVAP: Multicentre Proteomic Endotyping of Ventilator-associated Pneumonia
Acronym: ClusterVAP
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); NOVA Medical School (Other); Rigshospitalet, Denmark (Other); Karolinska University Hospital (Other); University Hospital, Limoges (Other); King's College Hospital NHS Trust (Other); Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-04564-01
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Ventilator Acquired Pneumonia; Mechanical Ventilation Complication
Keywords: VAP; endotyping; mini-BAL
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected ventilator-associated pneumonia: Adult ICU patients receiving mechanical ventilation who undergo bronchoalveolar lavage (BAL) or mini-BAL for clinical suspicion of lower respiratory tract infection. Residual BAL fluid will be analyzed using proteomic profiling to identify biological subgroups ("pneumoclusters"). No experimental intervention is administered; all patients receive standard care.

SUMMARY:
Ventilator-associated pneumonia (VAP) is a common and serious infection in patients receiving mechanical ventilation in intensive care units. Current diagnostic methods are imprecise, leading to unnecessary antibiotic use and delayed treatment. The ClusterVAP study aims to identify biologically and clinically distinct subgroups of patients with suspected VAP by analyzing proteins in bronchoalveolar lavage (BAL) fluid using advanced proteomic techniques. This multicentre observational study will enroll approximately 400 adult patients from intensive care units in Sweden, France, Portugal, Denmark, and the United Kingdom. BAL or mini-BAL samples collected for clinical reasons will be analyzed to define "pneumoclusters" and explore their association with patient outcomes. The study will also identify candidate biomarkers that could support future diagnostic tools. No experimental treatments are given; all patients receive standard care. Results may improve diagnostic accuracy and guide personalized treatment strategies for critically ill patients.

DETAILED DESCRIPTION:
ClusterVAP is an exploratory, observational, prospective, multicentre cross-sectional study designed to identify biologically and clinically distinct subgroups ("pneumoclusters") among patients with suspected ventilator-associated pneumonia (VAP). The study will enroll approximately 400 adult patients admitted to intensive care units in Sweden, France, Portugal, Denmark, and the United Kingdom who are receiving mechanical ventilation and undergo bronchoalveolar lavage (BAL) or mini-BAL for clinical reasons.

Residual BAL supernatant will be processed for proteomic analysis using liquid chromatography tandem mass spectrometry (LC-MS/MS). Unsupervised consensus clustering will be applied to proteomic data, alone and in combination with clinical and microbiological variables, to define pneumoclusters. These clusters will be characterized by clinical features, microbiology, and radiology, and compared for 30-day outcomes including mortality, ventilator-free days, antibiotic-free days, ICU-free days, and hospital-free days. Differential protein abundance analysis will be used to identify candidate biomarkers for pragmatic cluster assignment.

Data will be collected in electronic case report forms hosted in REDCap, with built-in quality checks. All data will be pseudonymized, and biological samples will be stored under controlled conditions for up to ten years for confirmatory analyses. No experimental interventions are administered; all patients receive standard care. The study has been approved by the Swedish Ethical Review Authority (Dnr 2025-04564-01) and equivalent bodies in participating countries. Results will be disseminated through peer-reviewed publications and scientific conferences, with statistical code shared for transparency.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years) admitted to an intensive care unit (ICU). Receiving invasive mechanical ventilation. Undergoing bronchoalveolar lavage (BAL) or mini-BAL on clinical indication for suspected lower respiratory tract infection.

New or worsening clinical signs compatible with lower respiratory tract infection within the preceding 24 hours, defined as the treating clinician's suspicion plus at least one of:

Body temperature >38 °C or <36 °C. Visually purulent tracheal secretions. Signs of reduced oxygenation (e.g., increased FiO₂ and/or decreased arterial pO₂, increased positive end-expiratory pressure or driving pressure).

Request for chest radiograph to investigate infection or new infiltrate. Initiation of antibiotic therapy targeting lower respiratory tract infection.

Exclusion Criteria:

BAL or mini-BAL performed solely for screening without suspicion of infection. Concurrent enrolment in the VAPmarkers study (reserved for external validation).

Age <18 years. Any condition that, in the opinion of the investigator, would preclude safe participation or confound study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted to intensive care units in Sweden, France, Portugal, Denmark, and the United Kingdom who are receiving invasive mechanical ventilation and undergo bronchoalveolar lavage (BAL) or mini-BAL for clinical suspicion of lower respiratory tract infection. Patients are enrolled at the time of sampling and followed for 30-day outcomes. No experimental interventions are administered; all patients receive standard care.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Distribution of patients into biologically distinct clusters ("pneumoclusters") based on BAL proteomic data | Day 0 (at enrolment)
  Unsupervised consensus clustering of bronchoalveolar lavage (BAL) proteomic profiles, alone and in combination with clinical and microbiological variables, will be performed to classify patients with suspected ventilator-associated pneumonia into biologically distinct clusters ("pneumoclusters"). The number of clusters, the number of patients per cluster, and key distinguishing features will be reported.

SECONDARY OUTCOMES:
30-day all-cause mortality | 30 days after enrolment
  Mortality status compared across identified clusters.
Ventilator-free days | 30 days after enrolment
  Number of days alive and free from invasive mechanical ventilation.
Antibiotic-free days | 30 days after enrolment
  Number of days alive and not receiving systemic antibiotics.
ICU-free days | 30 days after enrolment
  Number of days alive and not in an intensive care unit.
Hospital-free days | 30 days after enrolment
  Number of days alive and not hospitalized.

OTHER OUTCOMES:
Identification of candidate protein biomarkers for cluster assignment | Day 0 (at enrolment)
  Differential abundance analysis of bronchoalveolar lavage (BAL) proteomic data will be performed to identify candidate protein biomarkers that distinguish biologically defined patient clusters ("pneumoclusters"). The analysis will aim to derive a minimal set of proteins suitable for pragmatic cluster assignment in future cohorts. Results will include fold changes, statistical significance (e.g., adjusted p-values), and performance metrics (e.g., AUC) for each candidate biomarker.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be made available upon reasonable request to the corresponding author, subject to approval by relevant ethics committees and execution of appropriate data transfer agreements. Statistical code will be shared alongside the main publication. No genetic data will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available after publication of the main results and will remain available for up to 10 years after study completion or until the destruction of biological samples, whichever occurs first.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or healthcare institutions who submit a methodologically sound proposal. Requests should be directed to the corresponding author and will require approval by the study steering committee and relevant ethics committees.